CLINICAL TRIAL: NCT04992858
Title: A Phase II Study of the Ningetinib in Advanced NSCLC With MET Exon 14 Skipping Mutations
Brief Title: Ningetinib in Advanced NSCLC Skipping Mutations With MET Exon 14 Skipping Mutations
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT053-NSCLC-201
Record Dates: First submitted 2021-07-14; First posted 2021-08-05 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-07

CONDITIONS: Advanced NSCLC

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CT053PTSA (Experimental): 60 mg/d, starting on the first day
  Interventions: Drug: CT053PTSA

INTERVENTIONS:
Drug: CT053PTSA — CT053PTSA will be administered orally once a day
  Other Names: Ningetinib

SUMMARY:
This is a phase II, Single-arm,Open-label Study evaluating the safety and efficacy of CT053PTSA in Advanced Solid Tumors With MET Exon 14 Skipping Mutations

DETAILED DESCRIPTION:
This study is being carried out in two parts, part 1 and part 2. Part 1:Observation phase of dose tolerance: Objective To observe the tolerability and safety of 60 mg CT053PTSA in advanced NSCLC patients with Metex14 skipping mutation, and to determine the recommended dose (RED) in the dose expansion phase。 Part 2: This is the expansion part and will continue to evaluate the safety and efficacy of CT053PTSA at the dose of RED in advanced NSCLC patients with Metex14 skipping mutation.

ELIGIBILITY:
Inclusion Criteria:

* Age:18-75 years, male or female.
* Histologically or cytologically confirmed IIIB-IV- Advanced NSCLC
* There was a Metex 14 skipping mutation in plasma and / or tissue
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 ~2
* Life expectancy of greater than 12 weeks.
* Evaluable disease based on Response Evaluation Criteria In Solid Tumors (RECIST) 1.1
* Adequate organ function.
* Contraception, fertility and not lactating female subjects: screening blood pregnancy test must be negative
* Voluntarily join the study and sign informed consent ad has good compliance.

Exclusion Criteria:

* EGFR or ALK or ROS1 gene mutation was positive
* Anthracycline, nitrosourea, and mitomycin within 6 weeks; traditional Chinese medicine for anti-tumor within 2 weeks;other anti-tumor therapies within 4 weeks, Previously or currently participating in other clinical trials within 4 week, Prior therapies with c-MET targeted drugs; Had received vaccine within 4 weeks prior to study treatment or had a plan to receive vaccine during the trial.
* Not recovered from adverse events due to a previously administered agent.
* Symptomatic, untreated or unstable central nervous system metastases/ spinal cord compression, cancerous meningitis, or meningitis.
* Patients with other malignant tumors except NSCLC within 5 years before the first use of drugs do not include those with negligible risk of metastasis or death (such as expected 5-year OS > 90%) and expected to be cured after treatment, or any other tumors that have been cured (no evidence of recurrence within 5 years)
* There are prescribed cardiovascular and cerebrovascular risk factors
* Patients with evidence of bleeding tendency, or melena or hematemesis within 2 months; or visceral bleeding that may occur considered by investigator
* History of thyroid dysfunction, and the thyroid function cannot be maintained at the normal range with drugs.
* There are uncontrollable and active infections
* Uncontrollable massive pleural / ascites or pericardial effusion
* Clinically significant gastrointestinal abnormalities may affect the drug intake, transport or absorption (such as inability to swallow, chronic diarrhea, intestinal obstruction, etc.), or total gastrectomy subjects;
* a history of psychotropic drug abuse and can not quit or have mental disorders
* Any other reason the investigator considers the patient is not suitable to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-11-27 (Estimated); Primary Completion 2024-09-09 (Estimated); Study Completion 2024-12-09 (Estimated)

PRIMARY OUTCOMES:
Recommended Extended Dose | Cycle 1Day 1 to Cycle 1 Day 28±3
  Recommended dose for expansion phase
Objective response rate | up to 4 years
  Objective response rate (ORR) is defined as the percentage of the participants in the analysis population who have a confirmed complete response (CR) or partial response (PR) based on RECIST 1.1 by investigators

SECONDARY OUTCOMES:
Duration of response | up to 4 years
  Defined as the time from the earliest date of qualifying response until earliest date of disease progression, per RECIST v1.1, or death from any cause, whichever comes first. Includes participants with complete response or partial response
Progression-free survival | up to 4 years
  defined as the time from date of randomization until the earliest date of disease progression, as determined by independent central review of objective radiographic disease assessments per RECIST 1.1, or death from any cause, whichever comes first.
Overall survival | up to 4 years
  Defined as time from date of randomization to date of death due to any cause. OS was calculated using product-limit (Kaplan-Meier) method for censored data.
Disease Control Rate | up to 4 years
  proportion of patients with best overall response of CR, PR or stable disease (SD)
Adverse events related to CT053 | up to 4 years
  description, timing, grade (Common Terminology Criteria for Adverse Events Version 5.0 [CTCAE v5.0]), severity, seriousness, and relatedness

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, MD, Principal Investigator — Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: No